CLINICAL TRIAL: NCT06994390
Title: Neuropathic Pain Intervention With tDCS in Brazilian Military Personnel Randomized Controlled Trial
Brief Title: Neuropathic Pain Intervention With tDCS in Brazilian Military Personnel (NeuBRAIN Trial)
Acronym: NeuBRAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital da Polícia Militar de Goiás (Network)
Collaborators: Hospital das Clínicas de São Paulo - SP (Unknown)
Responsible Party: Principal Investigator, Eline Rozária Ferreira Barbosa, Principal Investigator, Hospital da Polícia Militar de Goiás
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NeuBRAIN RCT protocol
Record Dates: First submitted 2025-04-07; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Neuropathic Pain; Sleep Quality; Transcranial Direct Current Stimulation
Keywords: transcranial current stimulation; neuropathic pain; sleep
MeSH Terms: conditions — Neuralgia; Sleep Initiation and Maintenance Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The intervention will be carried out into two-weeks daily consecutive sessions of 20 minutes each, with 1 session/day, and a weekend interval. Direct current stimulation will be administered through an electrical stimulator model MicroEstim Genius (NKL), Brusque, Brazil. During the session, the participants will be awake and seated in a comfortable seat. The environment will be air-conditioned, free of visual and auditory stimuli.
  The sessions will be conducted by a trained health professional. The groups will receive single-phase direct current with an intensity of 2 mA up, according to data presented by Pacheco-Barrios et al. (2021). Electrodes with a size of 35cm² (5 x 7 centimeters) will be used. Electrodes will be placed on the scalp, fixed with elastic bands, and immersed in 10 to 12 mL of saline solution.
  The electrode montage will be performed for one of two possible targets: anodal stimulation over DLPFC or anodal stimulation over M1, and also sham in both targets.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A triple-blinding strategy will be implemented, including participants and outcome assessors, as well as staff responsible for recruitment and statistical analysis. To ensure proper intervention, only the health professional administering the treatment will know each participant's assigned group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anodal tdcs over the primary motor (M1) (Active Comparator): Anode placement will be positioned over M1, using the international 10-20 EEG system (C3/C4 for left or right M1).
  Cathode placement will be on the contralateral supraorbital area (above the eyebrow) to complete the circuit.
  Interventions: Device: tDCS
- Anodal tdcs over the dorsolateral prefrontal cortex (DLPFC) (Active Comparator): Anode placement positioned over dorsolateral prefrontal cortex (DLPFC), using the international 10-20 EEG system (F3/F4 for left or right DLPFC).
  Cathode placement will be on the contralateral supraorbital area (above the eyebrow) to complete the circuit.
  Interventions: Device: tDCS
- sham tdcs over M1 or DLPFC (Sham Comparator): The sham group will be divided in half of participants with Sham M1 and the other half as Sham DLPFC.
  Interventions: Device: sham intervention

INTERVENTIONS:
Device: tDCS — This group will receive single-phase direct current with an intensity of 2 mA up. Electrodes with a size of 35cm² (5 x 7 centimeters) will be used. Electrodes will be placed on the scalp, fixed with elastic bands, and immersed in 10 to 12 mL of saline solution.
  Other Names: transcranial direct current stimulation
  Arms: Anodal tdcs over the dorsolateral prefrontal cortex (DLPFC); Anodal tdcs over the primary motor (M1)
Device: sham intervention — The device displays will be identical across active and sham groups, and to ensure blinding, an active current will be applied for 30 seconds at the beginning and end of the sham stimulation to mimic the sensation of the current ramp experienced in active stimulation. Stimulations of less than 3 minutes of tDCS do not induce cortical excitability effects, according to Nitsche and Paulus (2000), being safely inactive for the expected results.
  Arms: sham tdcs over M1 or DLPFC

SUMMARY:
This project protocol investigates the efficacy of transcranial direct current stimulation (tDCS) in treating neuropathic pain and improving sleep quality among Brazilian military personnel. Given the high prevalence of chronic pain and sleep disturbances in this population, and the limitations of current pharmacological treatments, our randomized, triple-blinded, sham-controlled trial explores the potential of tDCS as a non-invasive therapeutic intervention. The results of this study could have a significant impact on improving the well-being and performance of military personnel, while also reducing healthcare costs associated with long-term medication use.

DETAILED DESCRIPTION:
The intervention will be carried out into two-weeks daily consecutive sessions of 20 minutes each, with 1 session per day, and a weekend interval. Direct current stimulation will be administered through an electrical stimulator model MicroEstim Genius (NKL), Brusque, Brazil. During the session, the participants will be awake and seated in a comfortable seat. The environment will be air-conditioned, free of visual and auditory stimuli.

The sessions will be conducted by a trained health professional. The groups will receive single-phase direct current with an intensity of 2 mA up, according to data presented by Pacheco-Barrios et al. (2021). Electrodes with a size of 35cm² (5 x 7 centimeters) will be used. Electrodes will be placed on the scalp, fixed with elastic bands, and immersed in 10 to 12 mL of saline solution.

The electrode montage will be performed for one of two possible targets: anodal stimulation over DLPFC or anodal stimulation over M1, and also sham in both targets according to the participants' designations after randomization to one of the three groups.

The device displays will be identical across active and sham groups, and to ensure blinding, an active current will be applied for 30 seconds at the beginning and end of the sham stimulation to mimic the sensation of the current ramp experienced in active stimulation. Stimulations of less than 3 minutes of tDCS do not induce cortical excitability effects, according to Nitsche and Paulus (2000), being safely inactive for the expected results.

ELIGIBILITY:
Inclusion criteria:

* Military personnel (active and veterans) with chronic pain due to central or peripheral neuropathy and poor sleep quality;
* Age over 18 years old;
* Defined chronic NeP according to current guidelines (ICD-10 codes OR DN-4);
* Pain with an average intensity score above 40/100 mm on a visual analogue scale (VAS);
* Medication stability (chronic pain, depression, anxiety, sleep) for at least six weeks;
* Patients with bad sleep quality identified by the Pittsburgh Sleep Quality Index (PSQI) of 5 or more who do not improve under conventional treatment.

Exclusion criteria:

* General contraindications for tDCS: past head trauma, current epilepsy, intracranial ferromagnetic components, pacemaker, implanted microprocessors (i.e., cochlear implants);
* Pregnancy;
* Known major psychiatric disorders (as assessed by the DSM-5, e.g., psychosis), history of substance abuse, or work litigation issues;
* History of chronic refractory migraines;
* Non-treated moderate to severe sleep apnea defined as apnea/hypopnea index greater than 15 events per hour in baseline polysomnography;
* Skin conditions such as psoriasis or eczema that involve the scalp (Thair et al, 2017);
* Cancer-related pain;
* BMI >35, due to increased reports of pain associated with increased BMI (Basem, et al., 2021; Stokes et al., 2020);
* Patients who do not sign informed consent or do not want to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity by VAS | at baseline, at the end of the ten-day treatment and at follow-up, three weeks post-intervention.
  The primary outcome is a reduction in pain intensity by at least 30% (Dworkim et al., 2004; Farrar et al 2001). It will be assessed using the 100 mm Visual Analogue Scale (VAS), which consists of straight lines 100 mm long indicating "no pain" on one end and "worst possible pain or most intense pain possible" on the other (Huskisson, 1974). The VAS is scored by measuring the distance from the "no pain" end of the line. Pain intensity will be assessed daily during the 10day intervention.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | It will be measured at baseline, at the end of the ten-day treatment and at follow-up, three weeks post-intervention.
  Before and after the interventions, sleep secondary outcomes will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which global score ranges from 0 to 21, with a higher score indicating poorer sleep quality. Each of the 7 component scores also range from 0 to 3, where a higher score on each component signifies more difficulty.
Epworth Sleepiness Scale (ESS) | at baseline, at the end of the ten-day treatment and at follow-up, three weeks post-intervention.
  Before and after the interventions, the Epworth Sleepiness Scale (ESS) will be applied. The ESS has a minimum score of 0 and a maximum score of 24. Higher scores indicate greater daytime sleepiness, with scores above 10 suggesting excessive daytime sleepiness. A higher score is therefore indicative of a worse outcome, as it signifies a greater tendency to fall asleep in various situations.
the Visual Analogue Scale for Fatigue Severity (VAS-F) | measured at baseline, at the end of the ten-day treatment and at follow-up, three weeks post-intervention.
  Before and after the interventions, we will apply the Visual Analogue Scale for Fatigue Severity (VAS-F). The VAS-F uses a 100 mm line and scores are determined by measuring the distance from one end of the line to the point the individual marks, resulting in a score between 0 and 100. A higher score indicates greater fatigue severity.
Polysomnographic evaluation - time | PSG will be measured at baseline and at the end of the ten-day treatment.
  Sleep evaluation with Type 2 polysomnography (PSG) will be recorded at baseline and will access time in bed (minutes), time to sleep onset (minutes), total sleep time (minutes), sleep latency (minutes), REM latency (minutes), wake after sleep onset (minutes).
Polysomnographic evaluation - arousal index | PSG will be measured at baseline and at the end of the ten-day treatment.
  The Arousal Index (AI) in polysomnography will be measured by counting the total number of arousals during sleep and dividing it by the total sleep time.
Polysomnographic evaluation - sleep efficiency | PSG will be measured at baseline, at the end of the ten-day treatment.
  Sleep efficiency (SE) will be calculated as the total sleep time (TST) divided by the total time in bed, multiplied by 100. A higher SE percentage indicates that more time in bed is spent actually sleeping. Normal sleep efficiency is generally considered to be 85% or higher.
Polysomnographic evaluation- sleep stages | at baseline, at the end of the ten-day treatment.
  Sleep stages will be scored by analyzing 30-second epochs of polysomnographic recordings using electroencephalogram (EEG), electrooculogram (EOG), and electromyogram (EMG) signals.
Polysomnographic evaluation- PLMI | PSG will be measured at baseline, at the end of the ten-day treatment.
  The Periodic Limb Movement Index (PLMI) is calculated as the number of periodic limb movements during sleep (PLMS) per hour of sleep time. According to the American Academy of Sleep Medicine (AASM) scoring criteria, a limb movement (LM) is scored if there is an increase in anterior tibialis electromyogram (EMG) activity of more than 8 microvolts above resting EMG, lasting between 0.5 to 10 seconds. Periodic limb movements (PLMS) are defined as a series of at least four consecutive limb movements, each separated by an inter-movement interval of 5 to 90 seconds. The PLMI is computed by dividing the total number of PLMS by the total sleep time in hours, yielding PLMS per hour of sleep (PLMS/h). A PLMI greater than 15 per hour in adults is considered clinically significant for periodic limb movement disorder.

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index Addendum for Posttraumatic Stress Disorder (PSQI-A) | at baseline and at the end of 10-day treatment
  A possible confounder to be controlled for will be assessed by the Pittsburgh Sleep Quality Index Addendum for Posttraumatic Stress Disorder (PSQI-A) addresses patients exposed to trauma and was validated in U.S. male military veterans (Insana et al., 2013) and also in Portuguese by Gonçalves and Lima (2014). Seven items assess the frequency of hot flashes; general nervousness; memories or nightmares of the traumatic experience; severe anxiety or panic, not related to traumatic memories; nightmares, not related to traumatic memories; episodes of terror or screaming during sleep without full awakening; and episodes of staged dreams (Germain et al., 2005).
  The PSQI-A (Pittsburgh Sleep Quality Index Addendum for Posttraumatic Stress Disorder) ranges from 0 to 21. Higher scores indicate a poorer outcome in PTSD symptom severity and a worse sleep quality. Scores of 5 or less generally indicate good sleep quality. Higher scores on the PSQI-A are also associated with more combat exposure.
the Depression-Anxiety-Stress Scales-21 (DASS-21) | at baseline and at the end of 10-day treatment
  Possible confounders to be controlled for will be assessed by the Depression-Anxiety-Stress Scales-21 (DASS-21) validated for Portuguese (Lovibond and Lovibond, 1995; Vignola and Tucci, 2014), that measures the levels of depression, anxiety and stress based on behaviors and feelings experienced in the last seven days. The DASS-21 has a score range from 0 to 63, in which the total score is calculated by summing the scores from all three subscales (depression, anxiety and stress). Higher scores indicate a more severe or frequent experience of depression, anxiety, and stress symptoms, i.e., a worse outcome.
Sociodemografic characteristics - DOB | at baseline
  The sociodemographic data collected will include date of birth (DD/MM/YYYY)
Sociodemografic characteristics - age | at baseline
  The sociodemographic data collected will include age (years)
Sociodemografic characteristics - educational level | at baseline
  The sociodemographic data collected will include educational level (length in years).
Sociodemografic characteristics - marital status | at baseline
  The sociodemographic data collected will include marital status (single, married, widow, other)
Sociodemografic characteristics - previous diseases | at baseline
  The sociodemographic data collected will include pre-existing diagnoses (name of the disease)
Sociodemografic characteristics - medication use | at baseline
  The sociodemographic data collected will include medication currently and previously used that may interfere with the results.
Sociodemografic characteristics- weight | at baseline
  Weight (kilograms) will be measured in a scale in the baseline.
sociodemografic characteristics- height | at baseline
  Height will be measured in centimeters with a height and weight scale, in which a sliding bar that is lowered to touch the top of the person's head, and the measurement is then read from the scale's markings. In addition, weight and height will be combined to report body mass index- BMI - in kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa Bueno, MD, PhD, Study Director — São Paulo University
Locations (1):
- Hospital da Polícia Militar de Goiás, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be available, after de-identification. There will be shared the study protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after one year of the publication of the main results (2030 March) - for 3 years.
Access Criteria: Data will be shared with researchers upon request for analyses related to the study's objectives, via a secure data repository.

REFERENCES:
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Mehta S, McIntyre A, Guy S, Teasell RW, Loh E. Effectiveness of transcranial direct current stimulation for the management of neuropathic pain after spinal cord injury: a meta-analysis. Spinal Cord. 2015 Nov;53(11):780-5. doi: 10.1038/sc.2015.118. Epub 2015 Jul 21. PMID 26193817
- [Background] Pacheco-Barrios K, Cardenas-Rojas A, Thibaut A, Costa B, Ferreira I, Caumo W, Fregni F. Methods and strategies of tDCS for the treatment of pain: current status and future directions. Expert Rev Med Devices. 2020 Sep;17(9):879-898. doi: 10.1080/17434440.2020.1816168. Epub 2020 Sep 15. PMID 32845195
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728